CLINICAL TRIAL: NCT03979118
Title: Exercise Prescription in Patients With Bone Metastases: Identifying Clinical Tools to Overcome Clinician Concerns Regarding Skeletal Related Events (Ex-Met Study)
Brief Title: Exercise Prescription in Patients With Bone Metastases
Acronym: Ex-Met
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Irish Cancer Society (Other); St. James's Hospital, Ireland (Other); Tallaght University Hospital (Other); Our Lady's Hospice & Care Services, Harold's Cross (Other)
Responsible Party: Principal Investigator, Emer Guinan, Principal Investigator, University of Dublin, Trinity College
Other Study IDs: PAL17GUI
Record Dates: First submitted 2019-05-29; First posted 2019-06-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Advanced Cancer; Bone Metastases
Keywords: Physical Activity; Skeletal Related Events
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer which has spread to the bone, causing bone metastases (bone tumours) can weaken bone health and increase risk of fractures (breaks). Consequently, patients can be unsure whether to exercise and health professionals can be unsure what exercise advice is suitable. Despite this, it is well known that exercise improves quality-of-life for patients with bone metastases and therefore it is important that exercise is prescribed to these patients.

This study aims to increase understanding of the link between daily exercise and risk of fracture in patients with bone metastases.

DETAILED DESCRIPTION:
It remains unclear if being physically active increases the risk of skeletal-related events in patients with bone metastases. Many health professionals report fracture risk as the primary concern with exercise prescription, despite a recognition of the importance of exercise participation. Consequently, health professionals can be hesitant to offer exercise advice and many patients are physically inactive. With increasing evidence supporting the benefits of exercise in metastatic bone disease, there is a need to address exercise-related concerns.

Clinical scoring systems such as Mirel's classification, are considered predictive of pathological fracture risk. While scoring algorithms have considerable potential to inform exercise eligibility in this population, to date the applicability of such clinical measures for exercise prescription have been inadequately studied. This study will examine the relationship between habitual physical activity, captured objectively by accelerometry, and skeletal related events (pathologic fracture, spinal cord compression, necessity for radiation to bone or surgery to bone pathological fracture) in patients with metastatic disease (n=100). Clinical data including fracture risk and Skeletal Related Events (SREs), Physical Activity (PA) data and subjective measures of pain, sleep, Quality of Life (QoL) and exercise barriers and benefits will be collected at baseline. Fracture risk will be determined at baseline using Mirel's Classification, which will be assessed by a radiologist affiliated with the study research team.

With treatment advances, patients with bone metastases secondary to advanced cancer are living longer. Consequently, optimising quality-of-life is a key priority and exercise has many recognised benefits in this domain. This research will explore the association between daily activity levels and skeletal complications in patients with bone metastases, by examining methods of identifying patients who are suitable to exercise, therefore improving exercise prescription practice and exercise participation safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bone metastases on radiological imaging as a result of breast, prostate or lung cancer.
* Initial systemic or local therapy post-diagnosis completed
* Commenced on bone modifying agents (BMAs)
* Provide signed and dated informed consent form

Exclusion Criteria:

* Cauda equina or metastatic spinal cord compression (MSCC)
* Pre-existing chronic pain (persistent or recurrent pain lasting longer than 3 months) due to orthopedic, rheumatology or fibromyalgia condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary breast and prostate cancers who have completed initial systemic or local treatment and have commenced on bone modifying agents (BMAs) will be invited to participate. With an overall study accrual target of n=100, monthly recruitment rates will be monitored and the recruitment strategy will be expanded if necessary, in response to a pre-defined set of accrual milestones.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Skeletal Related Events (SRE) | Baseline
  History of pathologic fracture (confirmed on imaging), metastatic spinal cord compression (MSCC), radiation to the bone (for pain or impending fracture), surgery to the bone or pain crisis (requiring intervention or escalation of analgesia)
Physical Activity | Baseline
  Physical activity will be assessed using the the ACTi Graph physical activity accelerometer.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Baseline
  The Brief Pain Inventory (BPI), a pain assessment tool that rapidly assesses the severity of pain and its impact on functioning in people living with cancer will be used to measure both the severity of pain (sensory dimension) and interference of pain in the patient's life (reactive dimension). Pain is rated on a scale of 0 (no interference) to 10 (interferes completely). The arithmetic mean of the four severity items is used as a measure of pain severity (mean severity score 0-40 with higher scores indicating higher pain severity). The arithmetic mean of the seven interference items is used as a measure of pain interference (0-70 with a higher score indicating higher levels of pain interference).
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Bone Mestastases 22(QLQ-BM22) | Baseline
  The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Bone Metastases 22 (QLQ-BM22) will be administered to measure quality of life. The QLQ-BM22 is a 22 item self-administered questionnaire that is divided into the following categories: Painful Sites (PS), Pain Characteristics (PC), Functional Interference (FI), and Psychosocial Aspects (PA). A high score for the symptom scales represents a high level of symptomatology or problems, whilst a high score for the functional scales represents a high level of functioning. All items are scaled from 1 (not at all) to 4 (very much), in which a higher score indicates greater distress in symptom scales while a higher score in functional scale indicates greater functional ability.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  The Pittsburgh Sleep Quality Index (PSQI), a self-report questionnaire will be used to assess sleep quality. The PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totalling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Exercise Benefits Barriers Scale (EBBS) | Baseline
  The Exercise Benefits / Barriers Scale (EBBS) will be used to measure perceived benefits of and perceived barriers to exercise. The overall perceived-benefits score is calculated by summing up the 29 benefit items, with higher values indicating greater perceived benefits. When the Benefits Scale is used alone, the score range is between 29 and 116. An overall perceived-barriers score is also calculated by summing the 14 barriers items, with higher values indicating greater perceived barriers. When the Barriers Scale is used alone, scores range between 14 and 56.
  The instrument is scored in its entirety or as two separate scales. Scores on the total instrument can range from 43 to 172. The higher the score, the more positively the individual perceives exercise.

OTHER OUTCOMES:
Mirel's Classification | Baseline
  At baseline, a Radiologist affiliated with the study will read the most recently available imaging and report in line with Mirel's classification, a proposed scoring system for diagnosing impending pathologic fractures. Mirel's classification system establishes fracture risk based on site of lesion, size of lesion, nature of lesion and subjective pain severity which provides a score between 4-12. Prophylactic fixation is indicated for a lesion with an overall score of 9 or greater. A lesion with an overall score of 7 or less can be managed using radiotherapy and drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Sheill, PhD, Study Director — University of Dublin, Trinity College; Lucy Balding, M.B.,MSc, Principal Investigator — St. James's Hospital and Our Lady's Hospice Harold's Cross; Ray McDermott, PhD, Principal Investigator — Tallaght University Hospital
Locations (1):
- St. James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided